CLINICAL TRIAL: NCT00874835
Title: Endothelial Graft Injector Versus Folding Forceps Insertion During Descemet's Stripping Endothelial Keratoplasty (DSEK)
Brief Title: Corneal Endothelium Delivery Instrument
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ocular Systems, Inc. (Industry)
Collaborators: Wake Forest University (Other)
Responsible Party: Kurt R. Weber, Ocular Systems, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endo33171
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Corneal Transplantation
Keywords: Endothelial Keratoplasty; EK; Descemet Stripping Endothelial Keratoplasty; Corneal Transplantation; Keratoplasty; DSEK; DSAEK

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: EndoSaver™ Corneal Endothelium Delivery Instrument — Efficacy of device to maintain function and integrity of corneal endothelial cells during insertion into the eye during keratoplasty.

SUMMARY:
The purpose of this study is to determine whether the surgical outcomes in patients undergoing Descemet's Stripping Endothelial Keratoplasty (DSEK) are improved with the use of an insertion device over the traditional forceps insertion method.

DETAILED DESCRIPTION:
Laboratory studies and clinical functionality tests have shown that the study device safely forms the tissue without creasing or folding. It allows the allograft tissue to safely pass into the anterior chamber without compression, crushing, or squeezing the endothelial cells.

The device provides continuous irrigation into the eye to prevent collapse of the anterior chamber during insertion. Our study will focus on the safety and efficacy of the novel instrument over the current method of insertion (forceps).

FDA has classified the device as Class I, Reserved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fuchs endothelial dystrophy or bullous keratopathy determined to need a corneal transplant for visual restoration.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
6-month post-operative endothelial cell density | 6-months post-operatively

SECONDARY OUTCOMES:
12-month post-operative endothelial cell density | 12-months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Walter, MD, Principal Investigator — Wake Forest University Eye Center
Locations (1):
- Wake Forest University Eye Center, Winston-Salem, North Carolina, United States